CLINICAL TRIAL: NCT04444570
Title: Continuous Glycemia Monitoring in Perioperative Period in Patients Undergoing Total Knee or Hip Arthroplasty: a Protocol of Observational Study
Brief Title: Continuous Glycemia Monitoring in Perioperative Period in Patients Undergoing Total Knee or Hip Arthroplasty
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Artur Stolarczyk, Head of the Department of Orthopedics and Rehabilitation, Medical University of Warsaw
Other Study IDs: Glycemia / WarsawMU
Record Dates: First submitted 2020-06-19; First posted 2020-06-23 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Osteoarthritis, Knee; Osteoarthritis, Hip; Hyperglycemia; Diabetes Mellitus, Type 2
Keywords: osteoarthritis; hip; knee; diabetes; glycemia
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip; Hyperglycemia; Diabetes Mellitus, Type 2; Osteoarthritis; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Control group: 14 days before the date of the surgery every participant will have implemented the device for continuous glycemia measurement (Dexcom)
  Interventions: Device: Continuous glycemia measuring device (Dexcom) implantation into the subcutaneous tissue
- Study group: Right after the surgery every participant will have implemented the device for continuous glycemia measurement (Dexcom). During standard control visit 14 days after the surgery for skin sutures removal the device will be taken out and data of whole period of time will be collected
  Interventions: Device: Continuous glycemia measuring device (Dexcom) implantation into the subcutaneous tissue

INTERVENTIONS:
Device: Continuous glycemia measuring device (Dexcom) implantation into the subcutaneous tissue — 14 days before the date of the surgery and after the surgery patient will have implemented the device for continuous glycemia measurement (Dexcom). During standard control visit 14 days after the surgery for skin sutures removal the device will be taken out and data of whole period of time will be collected

SUMMARY:
All across surgery specialties, wound or implant infections constitute rare, yet potentially severe complications of surgical procedure. It is considered, that glucose metabolism disorders, e.g. diabetes, are one of the main risk factors of such condition.

Aim of the study The aim of the study is a prospective evaluation of glucose blood level and its variability during 2 weeks before hospitalization and 2 weeks of postoperative period in patients, that will undergo elective orthopaedic surgeries, and its impact on number of cardiovascular and orthopaedic complications.

Materials and methods To this study, patients qualified for elective total knee or hip replacement in the single orthopedic center will be recruited. 100 patients will be included in this study. Every patient will be evaluated on the risk of developing diabetes mellitus in 10 years time and on the risk of death in 10 years due to the cardiovascular events. 14 days before procedure patients will have continuous glucose level measurement sensor implemented in subcutaneous tissue. After 14 days, during standard visit for stitches removal, the sensor will be removed and glycemia data will be collected. Next, patients will have their casual glucose blood level checked and surgery outcome, cardiovascular events or surgery complication risk evaluated in 3-, 6- and 12 month follow-up visits.

Expected benefits of the study Results of this study may allow to define impact of orthopaedic treatment on glycemia and possible necessity to modify treatment of hyperglycemia in perioperative period in patients with Diabetes Mellitus type 2 (DM2). Moreover it will allow to specify change of glucose levels and possibly implicating a need to monitor perioperative glycemia in patients without carbohydrate metabolism disorders. Additionally, the study will help to evaluate corelation between perioperative glucose blood level and the risk of cardiovascular events or surgical complications in 1-year after the procedure, which may decrease the risk of such incidents in the future (e.g. by adequate control and effective treatment of hyperglycemia), hence may result in reduction of mortality and lesser lowering of the quality of life in patients with DM2 or high risk of it.

DETAILED DESCRIPTION:
In every surgical subspeciality surgical site or implants infections are not common but potentially devastating for patients health. One of the most known risk factors of such state is glucose metabolism disorders. Such pathologies, containing diabetes mellitus, are considered one of the most epidemic health-related problems in XXI century.

Diabetes is a civilization disease, caused mainly by obesity, unhealthy eating habits and lack of physical activity. It was concerning about 108 million people in 1980, while in next 40 years this number grew 4-times and is expecting to reach almost 600 million people in 2035.

Total joint arthroplasty is considered the most effective way of treating the end-stage osteoarthritis of hip and knee joints. It is estimated that every year more that one million total joint replacements are performed in Europe. It is believed that our community is getting older and that is the reason why the number of total joint replacements will be growing, as well as patients expectations towards it. Even though total knee and hip replacement have wonderful outcome and are improving significantly patients life and its quality, there are several potential side effect that might lower patients limb function.

There were several studies confirming increased risk of surgical site or implants infections in patients undergoing total joint replacements such as knee or hip, who had perioperative poor glycemic control or had treated diabetes mellitus. However, there is lack of literature concerning analysis of continuous glycemia measurements before and after hospital stay. There are some promises that glycemic disturbances during postoperative period might also increase risk of cardiovascular events in this time and more frequent periods of hypoglycemia, which might result in higher risk of unconsciousness and falls. What is more higher cardiovascular risk is corelated with higher risk of disability and death.

Results of this research will allow to investigate influence of orthopedic surgery on glycemia and possible modifications of hyperglycemia treatment in perioperative period in patients with diabetes or glucose intolerance. What is more it will allow to investigate changes of glycemia in patients with normal glycemia metabolism, potentially protecting them from hypoglycemia during hospital stay and increasing their awareness of potentially suffering diabetes mellitus in the future. Additionally, this study will allow to corelate perioperative glycemia levels with risk of cardiovascular events in one year follow-up, and its influence on surgical site and implants complications. Thanks to these findings surgeons will be able to lower the risk of such complications in the future, hence lowering mortality and quality of life, especially in patients with diabetes mellitus and from the group with high risk of developing this disorder.

Nowadays, with technological development concerning our every day life, also devices used in medicine are getting more and more sophisticated and are making patients lifes easier. One of the most prominent examples of such device are the "discs" implanted into the subcutaneous tissue which might measure patients glycemia level. Thanks to it patients no longer need to measure it with traditional glucometers, which action relayed on blood samples collected from the tip of the finger. It was associated with every day unpleasant needling. Nowadays modern solution allow patients to get the result from their devices on their smartphones by only sliding it above the place of the implanted device.

Taking into considerations, such a wide spread of diabetes mellitus in our population it is obvious, that among patients qualified for total hip or knee arthroplasty many of them will have this disease. Adding to it common risk factors of diabetes and osteoarthritis, such as obesity, it seems that number of patients with such diseases is much bigger than it seems. According to the literature mentioned above it is obvious that microangiopathic changes, as well as hyperglycemia, have negative influence on wound healing, surgery itself and might increase the risk of periprosthetic infections. It is worthy to look for ways to optimize patients care in perioperative period.

Additional good side of this study is a fact, that it contains patients without recognized diabetes mellitus to assess their glycemia fluctuations, without carbohydrate metabolism disorders. Such knowledge might improve and allow to develop the algorithm of perioperative care for the high number of patients, who in such demanding for their body period are exposed to significant glycemia fluctuations.

What is more, it must be admitted that this study has unique model (described below), in which glycemia monitoring will contain both pre- and postoperative period of every included patient. Such way of analyzing patients allows to produce "perfect control group", because every measurements after the surgery has its counterpart before the surgery.

The aim of this project is to prospectively evaluate the level of glycemia and its variability in patients undergoing elective orthopedic surgeries during one month (two weeks before the surgery and two weeks postoperatively) and its influence on the number of cardiovascular and orthopedic complications. What is more the investigators want to evaluate its influence on objective functional outcome of the surgery in one year follow-up. It seems that long bone surgery as a stress factor might increase the risk of developing diabetes or glucose intolerance, what might increase the risk of cardiovascular diseases and number of complications.

To this prospective observational study, patients qualified for elective total knee or hip replacement in the Department of Orthopedics and Rehabilitation in Miedzyleski Specialist Hospital in Warsaw will be recruited. 100 patients will be included.

There were several studies confirming increased risk of surgical site or implants infections in patients undergoing total joint replacements such as knee or hip, who had perioperative poor glycemic control or had treated diabetes mellitus. However, there is lack of literature concerning analysis of continuous glycemia measurements before and after hospital stay. There are some premises that glycemic disturbances during postoperative period might also increase risk of cardiovascular events in this time and more frequent periods of hypoglycemia, which might result in higher risk of unconsciousness and falls. What is more higher cardiovascular risk is corelated with higher risk of disability and death.

Results of this research will allow to investigate influence of orthopedic surgery on glycemia and possible modifications of hyperglycemia treatment in perioperative period in patients with diabetes or glucose intolerance. What is more it will allow to investigate changes of glycemia in patients with normal glycemia metabolism, potentially protecting them from hypoglycemia during hospital stay and increasing their awareness of potentially suffering diabetes mellitus in the future. Additionally, this study will allow to corelate perioperative glycemia levels with risk of cardiovascular events in one year follow-up, and its influence on surgical site and implants complications. Thanks to these findings surgeons will be able to lower the risk of such complications in the future, hence lowering mortality and quality of life, especially in patients with diabetes mellitus and from the group with high risk of developing this disorder.

Nowadays, with technological development concerning our every day life, also devices used in medicine are getting more and more sophisticated and are making patients lifes easier. One of the most prominent examples of such device are the "discs" implanted into the subcutaneous tissue which might measure patients glycemia level. Thanks to it patients no longer need to measure it with traditional glucometers, which action relayed on blood samples collected from the tip of the finger. It was associated with every day unpleasant needling.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized in the Department of Orthopedics and Rehabilitation of Medical University of Warsaw
* Willingness to participate in the study
* Qualified for total knee or hip replacement due to the primary osteoarthritis
* Age above 18 years

Exclusion Criteria:

* No acceptance to participate in the study
* Qualified for non-surgical treatment
* Patients with other diseases but diabetes mellitus, compensated thyroid disorders and hypertension
* Patients with poorly-controled diabetes mellitus and/or poorly-controlled hypertension
* Patients with diabetes type 1
* Patients from the rest-home
* Patients who had previous lower limb surgeries
* Patients who in opinion of research team might be poorly compliant
* Patients during pregnancy
* Patients who are not fluent in polish language

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Power analysis was performed to assess how many patients should be included in the study. Determining effect size was hindered by lack of literature comparing mean values and standard deviations (SD) between groups with and without complications. The effect size can be deemed "large", described numerically as 0.8 by Cohen. However, we decide to be more conservative and used effect size of 0.6, located between "medium" and "large" in Cohen's scale. Standard p value of 0.05, beta value of 0.8 and allocation ratio of 1/1 were used, resulting in total needed sample size of 90 patients. Taking into consideration that 10 % of patients might drop off the follow-up predicted number of participants is 100.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Changes of glycemia levels during perioperative period | 4 weeks (14 days preoperatively and 14 postoperatively)
  Continuous glycemia level monitoring with use of subcutaneously implanted device
Rate and type cardiovascular events during follow-up | 12-months postoperatively
  Any cardiovascular events during follow-up (heart stroke, brain stroke, coronal arteries disease, transient ischaemic attack (TIA)
Rate and type of complications | 12-months postoperatively
  Any surgical site and/or implants complications during follow-up

SECONDARY OUTCOMES:
Objective functional outcome in Knee Injury and Osteoarthritis Outcome Score (KOOS) | 14-days, 3-, 6-, and 12- months postoperatively
  KOOS is a questionnaire designed to assess patient-relevant outcomes following knee injury. The KOOS assesses outcomes: pain, symptoms, activities of daily living, sport and recreation function, and knee-related quality of life. All items have five possible answer options scored from 0 (No problems) to 4 (Extreme problems). Scores between 0 and 100 represent the percentage of total possible score achieved.
Cardiovascular events and/or surgical site or implants complications | 12 months postoperatively
  Correlation of FINDRISC scale results with cardiovascular events and/or surgical site or implants complications

CONTACTS AND LOCATIONS:
Overall Officials: Artur Stolarczyk, qMD, PhD, Study Chair — Medical University of Warsaw

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Owens CD, Stoessel K. Surgical site infections: epidemiology, microbiology and prevention. J Hosp Infect. 2008 Nov;70 Suppl 2:3-10. doi: 10.1016/S0195-6701(08)60017-1. PMID 19022115
- [Background] de Oliveira AC, Sarmento Gama C. Surgical site infection prevention: An analysis of compliance with good practice in a teaching hospital. J Infect Prev. 2017 Nov;18(6):301-306. doi: 10.1177/1757177417703190. Epub 2017 Apr 27. PMID 29344100
- [Background] Ata A, Lee J, Bestle SL, Desemone J, Stain SC. Postoperative hyperglycemia and surgical site infection in general surgery patients. Arch Surg. 2010 Sep;145(9):858-64. doi: 10.1001/archsurg.2010.179. PMID 20855756
- [Background] Martin ET, Kaye KS, Knott C, Nguyen H, Santarossa M, Evans R, Bertran E, Jaber L. Diabetes and Risk of Surgical Site Infection: A Systematic Review and Meta-analysis. Infect Control Hosp Epidemiol. 2016 Jan;37(1):88-99. doi: 10.1017/ice.2015.249. Epub 2015 Oct 27. PMID 26503187
- [Background] Kharroubi AT, Darwish HM. Diabetes mellitus: The epidemic of the century. World J Diabetes. 2015 Jun 25;6(6):850-67. doi: 10.4239/wjd.v6.i6.850. PMID 26131326
- [Background] Skyler JS, Bakris GL, Bonifacio E, Darsow T, Eckel RH, Groop L, Groop PH, Handelsman Y, Insel RA, Mathieu C, McElvaine AT, Palmer JP, Pugliese A, Schatz DA, Sosenko JM, Wilding JP, Ratner RE. Differentiation of Diabetes by Pathophysiology, Natural History, and Prognosis. Diabetes. 2017 Feb;66(2):241-255. doi: 10.2337/db16-0806. Epub 2016 Dec 15. PMID 27980006
- [Background] Lubbeke A, Silman AJ, Barea C, Prieto-Alhambra D, Carr AJ. Mapping existing hip and knee replacement registries in Europe. Health Policy. 2018 May;122(5):548-557. doi: 10.1016/j.healthpol.2018.03.010. Epub 2018 Mar 17. PMID 29598886
- [Background] Pijls BG, Meessen JMTA, Tucker K, Stea S, Steenbergen L, Marie Fenstad A, Makela K, Cristian Stoica I, Goncharov M, Overgaard S, de la Torre JA, Lubbeke A, Rolfson O, Nelissen RGHH. MoM total hip replacements in Europe: a NORE report. EFORT Open Rev. 2019 Jun 3;4(6):423-429. doi: 10.1302/2058-5241.4.180078. eCollection 2019 Jun. PMID 31210979
- [Background] Ackerman IN, Dieppe PA, March LM, Roos EM, Nilsdotter AK, Brown GC, Sloan KE, Osborne RH. Variation in age and physical status prior to total knee and hip replacement surgery: a comparison of centers in Australia and Europe. Arthritis Rheum. 2009 Feb 15;61(2):166-73. doi: 10.1002/art.24215. PMID 19177522
- [Background] Kheir MM, Tan TL, Kheir M, Maltenfort MG, Chen AF. Postoperative Blood Glucose Levels Predict Infection After Total Joint Arthroplasty. J Bone Joint Surg Am. 2018 Aug 15;100(16):1423-1431. doi: 10.2106/JBJS.17.01316. PMID 30106824
- [Background] Maeda Y, Nakamura N, Tsujimoto T, Sugano N. Higher blood glucose and larger fluctuations detected postoperatively using continuous glucose monitoring: a preliminary study following total knee or hip arthroplasty. J Exp Orthop. 2019 Apr 1;6(1):15. doi: 10.1186/s40634-019-0181-9. PMID 30937670
- [Background] Kitsios K, Tsapas A, Karagianni P. Glycemia and cardiovascular risk: challenging evidence based medicine. Hippokratia. 2011 Jul;15(3):199-204. PMID 22435015
- [Background] Kishore P, Kim SH, Crandall JP. Glycemic control and cardiovascular disease: what's a doctor to do? Curr Diab Rep. 2012 Jun;12(3):255-64. doi: 10.1007/s11892-012-0268-5. PMID 22467273
- [Background] Brand-Miller J, Dickinson S, Barclay A, Celermajer D. The glycemic index and cardiovascular disease risk. Curr Atheroscler Rep. 2007 Dec;9(6):479-85. doi: 10.1007/s11883-007-0064-x. PMID 18377788
- [Background] Giorgino F, Leonardini A, Laviola L. Cardiovascular disease and glycemic control in type 2 diabetes: now that the dust is settling from large clinical trials. Ann N Y Acad Sci. 2013 Apr;1281(1):36-50. doi: 10.1111/nyas.12044. Epub 2013 Feb 6. PMID 23387439
- [Background] Lara-Pezzi E, Dopazo A, Manzanares M. Understanding cardiovascular disease: a journey through the genome (and what we found there). Dis Model Mech. 2012 Jul;5(4):434-43. doi: 10.1242/dmm.009787. PMID 22730474
- [Background] Mc Namara K, Alzubaidi H, Jackson JK. Cardiovascular disease as a leading cause of death: how are pharmacists getting involved? Integr Pharm Res Pract. 2019 Feb 4;8:1-11. doi: 10.2147/IPRP.S133088. eCollection 2019. PMID 30788283
- [Background] Vandersmissen GJ, Godderis L. Evaluation of the Finnish Diabetes Risk Score (FINDRISC) for diabetes screening in occupational health care. Int J Occup Med Environ Health. 2015;28(3):587-91. doi: 10.13075/ijomeh.1896.00407. PMID 26190733
- [Background] Bernabe-Ortiz A, Perel P, Miranda JJ, Smeeth L. Diagnostic accuracy of the Finnish Diabetes Risk Score (FINDRISC) for undiagnosed T2DM in Peruvian population. Prim Care Diabetes. 2018 Dec;12(6):517-525. doi: 10.1016/j.pcd.2018.07.015. Epub 2018 Aug 18. PMID 30131300
- [Background] Janghorbani M, Adineh H, Amini M. Evaluation of the Finnish Diabetes Risk Score (FINDRISC) as a screening tool for the metabolic syndrome. Rev Diabet Stud. 2013 Winter;10(4):283-92. doi: 10.1900/RDS.2013.10.283. Epub 2014 Feb 10. PMID 24841881
- [Background] Tomasik T, Krzyszton J, Dubas-Jakobczyk K, Kijowska V, Windak A. The systematic coronary risk evaluation (SCORE) for the prevention of cardiovascular diseases. Does evidence exist for its effectiveness? A systematic review. Acta Cardiol. 2017 Aug;72(4):370-379. doi: 10.1080/00015385.2017.1335052. Epub 2017 Jul 14. PMID 28705107
- [Background] Studzinski K, Tomasik T, Krzyszton J, Jozwiak J, Windak A. Effect of using cardiovascular risk scoring in routine risk assessment in primary prevention of cardiovascular disease: an overview of systematic reviews. BMC Cardiovasc Disord. 2019 Jan 9;19(1):11. doi: 10.1186/s12872-018-0990-2. PMID 30626326
- [Background] Dessein PH, Corrales A, Lopez-Mejias R, Solomon A, Woodiwiss AJ, Llorca J, Norton GR, Genre F, Blanco R, Pina T, Gonzalez-Juanatey C, Tsang L, Gonzalez-Gay MA. The Framingham Score and the Systematic Coronary Risk Evaluation at Low Cutoff Values Are Useful Surrogate Markers of High-risk Subclinical Atherosclerosis in Patients with Rheumatoid Arthritis. J Rheumatol. 2016 Mar;43(3):486-94. doi: 10.3899/jrheum.150510. Epub 2016 Jan 15. PMID 26773110
- [Background] Jorstad HT, Colkesen EB, Minneboo M, Peters RJ, Boekholdt SM, Tijssen JG, Wareham NJ, Khaw KT. The Systematic COronary Risk Evaluation (SCORE) in a large UK population: 10-year follow-up in the EPIC-Norfolk prospective population study. Eur J Prev Cardiol. 2015 Jan;22(1):119-26. doi: 10.1177/2047487313503609. Epub 2013 Sep 3. PMID 24002125
- [Background] Collins NJ, Prinsen CA, Christensen R, Bartels EM, Terwee CB, Roos EM. Knee Injury and Osteoarthritis Outcome Score (KOOS): systematic review and meta-analysis of measurement properties. Osteoarthritis Cartilage. 2016 Aug;24(8):1317-29. doi: 10.1016/j.joca.2016.03.010. Epub 2016 Mar 21. PMID 27012756
- [Background] Nilsdotter A, Bremander A. Measures of hip function and symptoms: Harris Hip Score (HHS), Hip Disability and Osteoarthritis Outcome Score (HOOS), Oxford Hip Score (OHS), Lequesne Index of Severity for Osteoarthritis of the Hip (LISOH), and American Academy of Orthopedic Surgeons (AAOS) Hip and Knee Questionnaire. Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S200-7. doi: 10.1002/acr.20549. No abstract available. PMID 22588745
- [Background] OECD (2017), "Hip and knee replacement", in Health at a Glance 2017: OECD Indicators, OECD Publishing, Paris.